CLINICAL TRIAL: NCT03216993
Title: The Shanghai Protocol for Early Enteral Nutrition in Mechanical Ventilated Patients
Brief Title: An Early Enteral Nutrition Protocol in Shanghai
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Erzhen Chen, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Shanghai EEN
Record Dates: First submitted 2017-07-08; First posted 2017-07-13 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Critical Illness; Enteral Feeding Intolerance
Keywords: feeding protocol
MeSH Terms: conditions — Critical Illness | interventions — Standard of Care; CARE protocol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Other): Standard care: patients receive enteral nutrition in accordance with the usual practice in the participating units
  Interventions: Other: Standard care
- Protocol care (Experimental): Protocol care： patient receive enteral nutrition in accordance with enteral nutrition protocol studied
  Interventions: Other: Protocol care

INTERVENTIONS:
Other: Standard care — Standard care: patients receive enteral nutrition in accordance with the usual practice in the participating units
  Arms: Standard care
Other: Protocol care — Protocol care： patient receive enteral nutrition in accordance with enteral nutrition protocol studied
  Arms: Protocol care

SUMMARY:
compare different enteral nutrition strategy in patients with mechanical ventilation

DETAILED DESCRIPTION:
There has been many evidence that deficiency in energy and protein take-in are associated with poor outcome in critical patients. To reach an adequate amount of energy and protein is critical in patients with respiratory failure and with mechanical ventilation, as it prevents muscle dystrophy and thus prevents ICU acquired weakness, leading to a better outcome in the end. Enteral Nutrition is preferred as it prevents gut dysfunction in respiratory failure patients, and may prevent further infection. But there are many challenge in implement a good enteral nutrition therapy, and energy or protein deficiency is common in patient with respiratory failure. There have been many protocols aiming at reaching enough enteral nutrition for ICU patients, most of which are based on a background of western and developed countries. The investigators developped a enteral nutrition protocol based on an unique cultural background of eastern developing country, trying to help the ICU patients reaching nutrition target, so that the patients may have better outcome.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients
* Receiving mechanical ventilation (MV) both Non-invasive ventilation and invasive ventilation
* Expecting MV more than 72 hours

Exclusion Criteria:

* Pregnancy
* ICU stay < 72hr

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
energy target fulfilling rate | 7 days from enrollment
  the proportion of patients in both arms meeting the targeted energy in-take
protein target fulfilling rate | 7 days from enrollment
  the proportion of patients in both arms meeting the targeted protein in-take

SECONDARY OUTCOMES:
mortality | 28 days from enrollment
  mortality

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Er Chen, Doctor, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No